CLINICAL TRIAL: NCT05868161
Title: Pounce™ Thrombectomy System Retrospective Registry
Acronym: PROWL
Status: Recruiting | Type: Observational
Sponsor: SurModics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SUR22-001
Record Dates: First submitted 2023-04-06; First posted 2023-05-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Arterial Disease; Acute Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Retrospective: All subjects in whom the Pounce Thrombectomy System was attempted will be included.
  Interventions: Device: Pounce Thrombectomy System

INTERVENTIONS:
Device: Pounce Thrombectomy System — Non-surgical removal of thrombi and emboli from the peripheral arterial vasculature with the Pounce Thrombectomy System.
  Other Names: Mechanical thrombectomy

SUMMARY:
The PROWL registry is an open-label retrospective, multi-center, US study of the Surmodics™ Pounce™ Thrombectomy System for the non-surgical removal of emboli and thrombi in the peripheral arterial vasculature.

ELIGIBILITY:
Inclusion Criteria:

* Subject underwent an endovascular intervention where the Pounce Thrombectomy System was attempted
* Subject is willing and able to provide informed consent prior to the collection of study data or a consent waiver is in place

Exclusion Criteria:

* Subject is under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects who have had an endovascular intervention where use of the Pounce Thrombectomy System was attempted
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Procedural Success | Peri-procedural (by the end of the index procedure)
  Restoration of pulsatile flow in the target lesion(s) with or without adjunctive treatment as determined by the core lab and physician
Incidence of device related Major Adverse Events (MAEs) | Procedure to 30 days
  Death, Unplanned major amputation (above ankle), Clinically Driven target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Technical success | Peri-procedural (by the end of the index procedure)
  Restoration of blood flow to the target lesion(s) with <50% residual thrombus without the need to initiate CDT or to proceed to open surgery or other endovascular thrombectomy device as determined by the core lab
Completeness of thromboemboli removal (by angiography) | Peri-procedural (by the end of the index procedure)
  Completeness of thromboemboli removal (by angiography) not including underlying atheroma as determined by the core lab and physician
Thrombo-aspiration in Peripheral Interventions (TIPI) flow rate | Peri-procedural (by the end of the index procedure)
  TIPI flow rate at the end of thrombectomy procedure and after any adjunctive procedures as determined by the core lab and physician.
Modified Society for Vascular Surgery (SVS) runoff | Pre-procedure, Peri-procedural (by the end of the index procedure)
  Pre-procedure vs. post-procedure runoff using a modified SVS runoff score as determined by the core lab and physician (if applicable).
Underlying atheroma stenosis | Peri-procedural (by the end of the index procedure)
  Length of underlying atheroma stenosis necessitating treatment compared to original lesion length as determined by the core lab and physician
Describe index procedural characteristics | Peri-procedural (by the end of the index procedure)
  Number of passes of Pounce Thrombectomy System
  * Total number of passes
  * Number of passes in each vessel
Adjunctive procedures | Peri-procedural (by the end of the index procedure)
  Percentage of subjects in whom adjunctive procedures were performed
  ▪ Treatment for: underlying atheroma, residual thrombus, residual embolus, other
Index procedure durations | Peri-procedural (by the end of the index procedure)
  Total procedure duration (minutes) Duration of Pounce Thrombectomy System use (minutes)
Characterize subject index procedure hospitalization course at discharge | Index procedure hospital admission to discharge, approximately 1 to 2 days
  Length of stay
Characterize subject index procedure hospitalization course at discharge | Index procedure hospital admission to discharge, approximately 1 to 2 days
  Time from end of procedure to discharge
Characterize subject index procedure hospitalization course at discharge | Index procedure hospital admission to discharge, approximately 1 to 2 days
  Incidence of same day discharge
Characterize subject index procedure hospitalization course at discharge | Index procedure hospital admission to discharge, approximately 1 to 2 days
  Incidence of next day discharge
Characterize subject index procedure hospitalization course at discharge | Index procedure hospital admission to discharge, approximately 1 to 2 days
  Incidence of ICU admission
Characterize subject index procedure hospitalization course at discharge | Index procedure hospital admission to discharge, approximately 1 to 2 days
  Duration of ICU admission
Primary vessel patency | 30 days
  Determined by the investigator using DUS or ABI
Rutherford class (if applicable) | Procedure to 30 days
  Improvement by at least one class at 30 days as compared to procedure
Rutherford classification (if applicable) | Baseline, at hospital discharge (approximately 1-2 days), 30 days
  Characterize Rutherford classification
Ankle Brachial Index (ABI) | Baseline to 30 days
  Change in ABI at 30 days compared to baseline.
Incidence of device related arterial AEs | 30 days
  Major bleeding (requiring transfusion) Arterial perforation Flow-limiting dissection (at the end of the procedure, prior to and following stenting, if performed) Distal embolization requiring surgical procedure or obstructing one of the major downstream vessels >70% (at the end of the procedure)
Incidence of all-cause: Death Unplanned major amputation (above ankle) Clinically driven TLR Clinically driven TVR | 30 days
Incidence of: Procedure-related SAEs Device-related (S)AEs | 30 days
Incidence of: Compartment syndrome requiring fasciotomy Major bleeding (requiring transfusion) unrelated to device | 30 days
Incidence of index procedure access site complications | 30 days
  Infection (requiring IV antibiotics or surgical treatment) Pseudoaneurysm (requiring surgical or endovascular treatment) Seroma (requiring surgical treatment) Other access site related AEs
  * Numbness
  * Other

CONTACTS AND LOCATIONS:
Overall Officials: Sean Lyden, MD, Principal Investigator — The Cleveland Clinic; Joseph Campbell, MD, Principal Investigator — OhioHealth
Locations (9):
- United States (9):
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Community Hospital, Munster, Indiana
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Allina Health, Minneapolis, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - Prisma Health Upstate, Greenville, South Carolina
  - North Central Heart, Sioux Falls, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Ascension Seton, Austin, Texas